CLINICAL TRIAL: NCT04431869
Title: In-Utero Vascular Accidents in Neonates From COVID-19 Infected Mothers
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1399
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Related; COVID; Intestinal Atresia; Limb Anomaly
MeSH Terms: conditions — Intestinal Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Mothers of children enrolled in the study with intestinal atresias or limb anomalies will undergo SARS-CoV-2 antibody testing to identify the possibility of asymptomatic carriers which may have occurred during the pregnancy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mothers that contract SARS-CoV-2 during pregnancy: To evaluate evidence for in-utero vascular accidents that may manifest as intestinal atresias and limb abnormalities in the first 30 days of life as well as rates of preterm labor, fetal growth restriction and spontaneous abortions in pregnant females that contract the SARS-CoV-2 virus during gestation.
  A multidisciplinary approach in conjunction with maternal fetal medicine (MFM), neonatology, and pathology will identify, and recruit infants whom were exposed to COVID-19 while in-utereo. This project will run in parallel with the institution's COVID-19 in Pregnancy Biobank that intends to obtain needed epidemiological and clinical data linked to biosamples to provide insight into SARS-CoV-2 in pregnant women and their infants. This study will request access to enrolled women infected during gestation and their neonates to assess for the conditions suggestive of in-utero vascular accidents such as intestinal atresias or limb anomalies.
- Infants noted to have intestinal atresias or limb anomalies: To evaluate children identified in the neonatal intensive care unit (NICU) as having evidence of intestinal atresias or limb anomalies for potential asymptomatic carriers of COVID-19 that could have contracted the disease during the pregnancy.
  Mothers of children identified will undergo SARS-CoV-2 antibody testing to identify the possibility of asymptomatic carriers which may have occurred during the pregnancy.

SUMMARY:
The pregnancy related pro-thrombotic state, in addition to the COVID-19 associated hypercoagulability may have unknown consequences to the developing fetus. Hence, this proposal seeks to address this question that may have important implications for women that contract this virus during gestation.

DETAILED DESCRIPTION:
Hypercoagulability and increased risk for venous thromboembolism (VTE) in severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infected patients are well documented in the growing body of literature, leading to institutional recommendations for daily pharmacologic anticoagulation while hospitalized and after discharge for some. While some of these hospitalized patients with COVID-19 infections have included pregnant women that also require inpatient pharmacologic anticoagulation and occasionally extended anticoagulation after discharge, little is known about the effects of the hypercoagulable COVID-19 induced state on the developing embryo, nor the necessary anticoagulation recommendation guidelines for these expecting mothers.

The pregnancy related pro-thrombotic state, in addition to the COVID-19 associated hypercoagulability may have unknown consequences to the developing fetus. Hence, this proposal seeks to address this question that may have important implications for women that contract this virus during gestation through the following specific aims.

Specific Aim 1: To evaluate evidence for in-utero vascular accidents that may manifest as intestinal atresias and limb abnormalities in the first 30 days of life as well as rates of preterm labor, fetal growth restriction and spontaneous abortions in pregnant females that contract the SARS-CoV-2 virus during gestation.

Rationale: Pregnancy produces a hypercoagulable state, this study intends to expand on the body of literature for COVID-19 manifestations by evaluating the additional virus-induced hypercoagulability on the developing embryo.

Methods: A multidisciplinary approach in conjunction with maternal fetal medicine (MFM), neonatology, and pathology, the study will identify, and recruit infants whom were exposed to COVID-19 while in-utereo. This project will run in parallel with the institution's COVID-19 in Pregnancy Biobank that intends to obtain needed epidemiological and clinical data linked to biosamples to provide insight into SARS-CoV-2 in pregnant women and their infants.

Specific Aim 2: To evaluate children identified in the neonatal intensive care unit (NICU) as having evidence of intestinal atresias or limb anomalies for potential asymptomatic carriers of COVID-19 that could have contracted the disease during the pregnancy.

Rationale: As high as 81% of patients that contract SARS-CoV-2 are asymptomatic or minimally symptomatic during the infection period. The long-term manifestation of the virus in these asymptomatic carriers, especially in pregnant women and their developing embryos, are presently unknown.

Methods: Mothers of children identified will undergo SARS-CoV-2 antibody testing to identify the possibility of asymptomatic carriers which may have occurred during the pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant females, 18 years and higher, with documented COVID-19 infection (antigen, PRC, or antibodies in a biologic sample) during gestation who received medical care at the University of Colorado Hospital (UCH) or Children's Hospital Colorado (CHCO)
* Neonates born to COVID-19 infected mothers
* Neonates ages 1-60 days of life with documented limb anomalies and intestinal atresias

Exclusion Criteria:

* Mothers with a history of vasoactive drug usage during pregnancy
* Mothers taking known teratogens during pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant females with documented COVID-19 gestational infections and their infants will be enrolled. Additionally, neonates with limb anomalies and intestinal atresias will be identified in the NICU and both infant and mother enrolled to identify if maternal SARS-CoV-2 infection occurred during the pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Rates of intestinal atresias and limb abnormalities | 12 months
  Evaluate rates of intestinal atresias and limb anomalies in neonates born to women that contract SARS-CoV-2 during pregnancy in the first 30 days of life
Rates of preterm labor, fetal growth restriction and spontaneous abortions | 12 months
  Rates of preterm labor, fetal growth restriction and spontaneous abortions for women that are known to be infected with SARS-CoV-2 during gestation
Rates of maternal SARS-CoV-2 infection among mothers to infants born with intestinal atresias or limb anomalies | 12 months
  For neonates identified in the NICU with intestinal atresias and limb anomalies, we will test the mothers for the presence of SARS-CoV-2 antibodies that may represent an asymptomatic carrier during gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study seeks to find a correlation between maternal COVID-19 infection and in-utero vascular accidents affecting the developing fetus. The knowledge gained from this multidisciplinary study may serve as the foundation for larger epidemiological studies that may query the longitudinal effects of this infection in mothers who contract the disease during pregnancy, as well as for their neonates. On a larger scale, if the study hypothesis is supported by the data, this may provide the foundation for future anticoagulation guidelines that may be enacted on certain women during gestation.